CLINICAL TRIAL: NCT05445999
Title: A Preliminary Study of Model-driven Individualized Transcranial Electrical Stimulation for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMHC-ISM-001
Record Dates: First submitted 2022-06-28; First posted 2022-07-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Insomnia
Keywords: Transcranial electrical stimulation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tES treatment (Experimental): Patients will receive ten sessions of daily individualized tDCS over a two-week period, delivered for 20 min at SMHC (sessions 2-11).
  Interventions: Device: High-Definition transcranial electrical stimulation

INTERVENTIONS:
Device: High-Definition transcranial electrical stimulation — The first and final sessions will include clinical assessments and acquisition of MRI and EEG data. To minimize variability, each patient will undergo tDCS at a consistent time in the afternoon or evening and will remain lying in bed with eyes closed throughout stimulation. Stimulation will be delivered using the GTEN 200 system (Magstim EGI, Oregon, USA), which also enables simultaneous EEG recording. The stimulation current will be limited to 1.5 mA, with a maximum of 0.15 mA per electrode (up to 20 electrodes). Electrode placement and current intensity will be individualized to achieve the targeted electric field strength (0.1 or 0.2 V/m at SMHC;). Each session will include 5 min of resting-state EEG immediately before and after stimulation to assess tDCS-induced changes in brain dynamics. Current onset and offset will be gradual, with 2-s ramp-up and ramp-down periods.

SUMMARY:
This study is designed to evaluate the efficacy and to explore the best individualized stimulus paradigm of transcranial Electrical Stimulation for insomnia patients.

DETAILED DESCRIPTION:
This study is an open-label clinical trial. A total of 40 patients with insomnia who meet the inclusion and exclusion of criteria will be recruited from the SMHC (20) and be assigned to receive individualized tDCS treatment. Patients will undergo ten days of daily individualized tDCS treatment for 20 min (sessions 2-11, SMHC) over a two-week period, which session 7 of patients for re-screening of tDCS target. In addition, normal control subjects and insomnia patients meeting eligibility criteria will be recruited from SMHC to identify biomarkers of wakefulness and sleep through simultaneous fMRI-EEG and high-density EEG recordings. These participants will not receive tDCS and will serve as controls for comparison with the treatment group.

ELIGIBILITY:
Participants will be recruited from the Shanghai Mental Health Center (SMHC) in Shanghai. Eligible insomnia participants were adults (18-50 years at SMHC) and diagnosed with insomnia disorder according to DSM-5 criteria by neurologists or psychiatrists using the procedure of Mini-International Neuropsychiatric Interview. Inclusion criteria were: (1) ≥ 9 years of education, (2) medication-free or had received stable medication for at least 2 months before entering the study and continued the same medication throughout the study. Exclusion criteria included: (1) serious medical, neurological, or psychiatric disorders other than anxiety or mild-to-moderate depression secondary to insomnia, (2) obstructive sleep apnea syndrome, (3) pregnancy or recent preparation for pregnancy, (4) previous treatments with ECT, rTMS, tES, and CBT-I.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | At baseline (prior to treatment), after 10 days of treatment ("post-treatment", week 2) and follow-up periods (weeks 3 and week 6, SMHC)
  The primary outcome is measured as the Insomnia Severity Index (ISI) at baseline (prior to treatment), after 10 days of treatment ("post-treatment", week 2) and follow-up periods (weeks 3 and week 6, SMHC).

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | At baseline (prior to treatment), after 10 days of treatment ("post-treatment", week 2) and follow-up periods (weeks 3 and week 6)
  Pittsburgh Sleep Quality Index (PSQI)
Change in Beck Depression Inventory, BDI | At baseline (prior to treatment), after 10 days of treatment ("post-treatment", week 2) and follow-up periods (weeks 3 and week 6)
  It consists of 21 items and uses a 0 to 3 severity scale. Total scores range from 0 to 63, with higher scores indicating more severe depression symptoms.
Change in Beck Anxiety Inventory, BAI | At baseline (prior to treatment), after 10 days of treatment ("post-treatment", week 2) and follow-up periods (weeks 3 and week 6)
  It is an inventory of anxiety symptoms with 18 items that are rated on a 5-point Likert scale(0 to 4). Total scores range from 0 to 72, with higher scores indicating more severe anxiety symptoms.
Change in Side-effect questionnaire | At baseline (prior to treatment), after 10 days of treatment ("post-treatment", week 2) and follow-up periods (weeks 3 and week 6).
  It consists of 10-item and uses 0 to 3 severity scale to rate the intensity of side effects. Total scores range from 0 to 30, with higher scores indicating more severe side-effect. It also assesses the relation between side-effect and the effects of tDCS using 0 to 4 scale. Total scores range from 0 to 40, with higher score indicating the greater relation.
sleep Diary | At baseline (prior to treatment), after 10 days of treatment ("post-treatment", week 2) and follow-up periods (weeks 3)
  A daily record of sleep-wake times and related lifestyle factors, such as caffeine intake, naps, and exercise, used to identify patterns and improve sleep
Remission Rate | week 2, weeks 3 and week 6
  Defined as ISI<8 based on the previous study

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD,MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China